CLINICAL TRIAL: NCT04052386
Title: Brief Alcohol Screening for Community College Students (BASICCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christine Lee, Research Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 50262; R34AA023047 (NIH)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Alcohol; Use, Problem
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions (BASICCS and assessment-only control group).
Who Masked: Participant
Masking Description: Participants were randomized into one of two conditions (BASICCS intervention and control [assessment-only]).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASICCS (Experimental): Participants randomized to the BASICCS condition received a personalized feedback intervention conducted through a web-conferencing platform. They also received up to 24 text messages with protective behavioral strategies for drinking during the following month.
  Interventions: Behavioral: BASICCS
- Control (No Intervention): Participants randomized to the control group did not receive any intervention. They were an assessment-only control group.

INTERVENTIONS:
Behavioral: BASICCS — Participants randomized to the BASICCS condition received a personalized feedback intervention conducted through a web-conferencing platform. The personalized feedback intervention included tailored feedback on drinking quantity and frequency of alcohol, BAC, alcohol-related consequences, normative perceptions of peer drinking, alcohol outcome expectancies, family history of risk, and financial costs of alcohol. They also received up to 24 text messages with protective behavioral strategies for drinking during the following month.
  Arms: BASICCS

SUMMARY:
The present study focuses on examining the feasibility, acceptability, and preliminary effects of an adapted alcohol intervention for high-risk college students attending community colleges. Investigators adapted BASICS (an efficacious in-person intervention developed for high-risk drinkers attending 4-year colleges and universities) to a web-conferencing format that allows the facilitator and participant to see and discuss live web-based personalized feedback. SMS text messages with protective behavioral strategies were also provided. The objective of the R34 was to establish feasibility and acceptability as well as to determine preliminary or likely effect sizes.

DETAILED DESCRIPTION:
Young adulthood (ages 18-29) is associated with increased risk for alcohol-related negative consequences; however, little is known about effective interventions for young adults attending community colleges (CCs). Thus, it is critical to develop an intervention that meets the various needs and demanding lifestyles of CC students. The investigators proposed to develop a user-friendly and convenient intervention that addresses relevant social norms, the impact of high-risk alcohol use on health and well-being in relevant life domains beyond student life and academic achievement, and provides ongoing exposure to behavior change strategies. To address the notable differences between CC students and traditional 4-year students, the investigators adapted BASICS to a web-conferencing format that allows the facilitator and participant to see and discuss live web-based personalized feedback (FB). This intervention for CC students, BASICCS, will focus on relevant normative feedback and alcohol's impact on multiple roles and personal goals of the CC student. Providing tips and protective behavioral strategies (PBS) after BASICS interventions via handouts or mailed postcards is standard practice and with preliminary evidence supporting the use of mobile phone text messaging (TM) or short message service (SMS) to reduce heavy-episodic drinking; thus, in this study SMS text messages were used to deliver ongoing protective behavioral strategies (PBS) the month after participating in the BASICCS session. The objective of this research was to establish feasibility and acceptability as well as to determine preliminary or likely effect sizes. CC student drinkers were recruited to participate and if eligible, they were randomized to one of two conditions (BASICCS or assessment-only control) and completed 1- and 3-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* being 18-29 years old; enrolled full- or part-time at one of the three community colleges where data collection took place; consuming 4+/5+ drinks for women/men on one occasion in the past month or exceeding weekly NIAAA drinking recommendations (8+/15+ for women/men); and possessing a cell phone with text-messaging capability

Exclusion Criteria:

* not meeting inclusion criteria, not consenting to participate

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | 1-month
  Number of standard drinks consumed each day of typical week past month
Daily Drinking Questionnaire | 3-month
  Number of standard drinks consumed each day of typical week past month
Frequency of Binge Drinking | 1-month
  Number of times in past month engaged in heavy episodic drinking (4+ drinks for women, 5+ drinks for men)
Frequency of Binge Drinking | 3-month
  Number of times in past month engaged in heavy episodic drinking (4+ drinks for women, 5+ drinks for men)
Estimated Blood Alcohol Concentration (eBAC) | 1-month
  estimated peak blood alcohol concentration
Estimated Blood Alcohol Concentration (eBAC) | 3-month
  estimated peak blood alcohol concentration
Brief Young Adult Alcohol Consequences Questionnaire | 1-month
  Number of alcohol-related consequences endorsed
Brief Young Adult Alcohol Consequences Questionnaire | 3-month
  Number of alcohol-related consequences endorsed

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Lee, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share limited datasets for the purposes of data analysis and dissemination.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data dictionaries and limited datasets can be made available starting in September 2020.
Access Criteria: Individual requests to access data with intended purpose should be made to Dr. Lee and will be reviewed by the investigative team.